CLINICAL TRIAL: NCT03883477
Title: Endoscopic Trigger Finger Release
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cedars-Sinai Medical Center (Other)
Responsible Party: Principal Investigator, David Kulber, MD, Principal Investigator, Cedars-Sinai Medical Center
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Pro00054088
Record Dates: First submitted 2019-03-15; First posted 2019-03-21 (Actual); Results first posted 2022-05-11 (Actual); Last update posted 2022-05-11 (Actual); Status verified 2022-04

CONDITIONS: Trigger Finger
Keywords: Tendinopathy; Trigger Finger
MeSH Terms: conditions — Trigger Finger Disorder; Tendinopathy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Endoscopic Release (Experimental): 12 patients recommended for surgical treatment of trigger finger will undergo endoscopic release.
  Interventions: Device: Endoscopic Release
- Standard Open Release (Active Comparator): 12 patients recommended for surgical treatment of trigger finger will undergo standard open surgical release.
  Interventions: Procedure: Standard Open Release

INTERVENTIONS:
Device: Endoscopic Release — Retrograde endoscopic release of the A1 pulley for treatment of trigger finger will be performed using a commercially available device by A.M. Surgical, Inc. This device has been cleared for marketing, sale and use by the U.S. Food and Drug Administration (FDA) for use as an Orthopedic manual surgical instrument based on its similarity in structure and function to previously used devices.
  Arms: Endoscopic Release
Procedure: Standard Open Release — Standard open surgical release of the A1 pulley for treatment of trigger finger.
  Arms: Standard Open Release

SUMMARY:
The purpose of this study is to compare recovery, scar, and patient satisfaction after retrograde endoscopic trigger finger release versus the standard open surgical treatment.

DETAILED DESCRIPTION:
Consecutive patients presenting with trigger finger interested in surgical release of the A1 pulley will be prospectively treated with endoscopic versus open surgical release of the A1 pulley. Study measures will include scar assessment based on the Patient and Observer Scar Assessment Scale (POSAS) administered at 1 week, 1 month, and 6 months post-operatively, overall satisfaction (scale of 1 to 10), days before return to work, duration of post-operative occupational therapy, pain medication use, operative time, and complication and recurrence rates.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years old
* Trigger finger diagnosis, recommended for surgical release
* Be in good health other than the trigger finger
* Have realistic expectations of surgical results
* Be willing to undergo surgical or endoscopic treatment
* Understand and be willing to follow all aspects of the study protocol and have signed and dated the Informed Consent Form and the Authorization for Use and Release of Health and Research Study Information (HIPAA) form prior to any study-related procedures being performed

Exclusion Criteria:

* Collagen-vascular, connective tissue, or bleeding disorder
* Pregnancy
* Regional sympathetic dystrophy
* Abscess or infection at time of planned surgery
* Have a condition or be in a situation that, in the Investigator's opinion, may put the subject at significant risk, may confound the study results, or may interfere significantly with the subject's participation in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2019-03-13 (Actual); Primary Completion 2021-09-24 (Actual); Study Completion 2021-09-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David A Kulber, MD, Principal Investigator — Cedars-Sinai Medical Center
Locations (1):
- Cedars-Sinai Department of Orthopedic Surgery, Los Angeles, California, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Endoscopic Release: 13 patients recommended for surgical treatment of trigger finger will undergo endoscopic release.
  Endoscopic Release: Retrograde endoscopic release of the A1 pulley for treatment of trigger finger will be performed using a commercially available device by A.M. Surgical, Inc. This device has been cleared for marketing, sale and use by the U.S. Food and Drug Administration (FDA) for use as an Orthopedic manual surgical instrument based on its similarity in structure and function to previously used devices.
- Standard Open Release: 13 patients recommended for surgical treatment of trigger finger will undergo standard open surgical release.
  Standard Open Release: Standard open surgical release of the A1 pulley for treatment of trigger finger.
Period: Overall Study
Arm/Group | Endoscopic Release | Standard Open Release
Started | 13 | 13
Completed | 12 | 12
Not Completed | 1 | 1
Not completed — Death | 1 | 0
Not completed — Protocol Violation | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Endoscopic Release | Standard Open Release | Total
Number analyzed (Participants) | 13 | 13 | 26
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 6 | 8 | 14
  >=65 years | 7 | 5 | 12
Age, Continuous [Mean (Standard Deviation); unit: years] | 65.53 (14.25) | 63.59 (10.66) | 64.55 (12.36)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 7 | 13
  Male | 7 | 6 | 13
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Scar Comparison Between Treatment Arms, as Measured by the Patient and Observer Scar Assessment Scale (POSAS)
Description: Questionnaires, completed by both the patient and the patient's surgeon/Physician Assistant (PA-C), contain 6 items on a 10-point scale (1 is best, 10 is worst). Scores range from 12 to 120 with 12 indicating normal skin and 120 indicating worst scar imaginable.
Time Frame: 1 Week, 1 Month and 6 Months after surgery
Population: One patient in the Endoscopic Release group died from causes unrelated to the study and one patient in the Standard Open Release treatment arm did not complete the first post-operative survey. All subjects were included in the final statistical analysis.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Endoscopic Release | Standard Open Release
Number analyzed (Participants) | 13 | 13
score on a scale
  1-Week Post-op: number analyzed (Participants) | 13 | 12
  1-Week Post-op | 27.2 (10.6) | 45.0 (19.8)
  1-Month Post-op | 31.2 (19.5) | 44.8 (13.1)
  6-Months Post-op: number analyzed (Participants) | 12 | 13
  6-Months Post-op | 16.8 (6.7) | 18.3 (8.1)
Statistical Analysis 1: Comparison: Endoscopic Release vs Standard Open Release; Test type: Other — The trial was powered to detect a difference in POSAS score of 10, deemed to be clinically significant by the investigators. To detect a mean difference in POSAS score of 10 points (SD = 8) with a two-sided significance level of 5% and power of 80% with equal allocation to two arms required 12 patients in each arm of the trial; p = 0.013, Wilcoxon (Mann-Whitney) — 1 week P-value
Statistical Analysis 2: Comparison: Endoscopic Release vs Standard Open Release; The trial was powered to detect a difference in POSAS score of 10, deemed to be clinically significant by the investigators. To detect a mean difference in POSAS score of 10 points (SD = 8) with a two-sided significance level of 5% and power of 80% with equal allocation to two arms required 12 patients in each arm of the trial; Test type: Other; p = 0.007, Wilcoxon (Mann-Whitney) — 1 month P-value
Statistical Analysis 3: Comparison: Endoscopic Release vs Standard Open Release; [analysis description as in outcome 1, analysis 2]; Test type: Other; p = 0.804, Wilcoxon (Mann-Whitney) — 6 month P-value

2. Secondary Outcome: Overall Patient Satisfaction: 10 Point Scale
Description: The patient's overall satisfaction after surgery based on a 10 point scale with 1 indicating no satisfaction and 10 indicating extremely satisfied.
Time Frame: End of Study (6 months after treatment)
Population: All available values included in the analysis.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Endoscopic Release | Standard Open Release
Number analyzed (Participants) | 12 | 9
score on a scale | 9.2 (2.6) | 8.2 (3.0)
Statistical Analysis 1: Comparison: Endoscopic Release vs Standard Open Release; Test type: Other; p = 0.142, Wilcoxon (Mann-Whitney)

3. Secondary Outcome: Weeks Before Return to Work
Description: Number of weeks after surgery before patient returns to work
Time Frame: End of study (6 months after treatment)
Population: All available values included. Not applicable for retired patients.
Measure: Mean (Standard Deviation); unit: Weeks
Arm/Group | Endoscopic Release | Standard Open Release
Number analyzed (Participants) | 9 | 8
Weeks | 2.6 (3.0) | 4.4 (5.7)
Statistical Analysis 1: Comparison: Endoscopic Release vs Standard Open Release; Test type: Other; p = 0.561, Wilcoxon (Mann-Whitney)

4. Secondary Outcome: Duration of Post-operative Therapy
Description: Number of days after surgery the patient participates in occupational therapy
Time Frame: End of study (6 months after treatment)
Population: All available data included in the analysis.
Measure: Mean (Standard Deviation); unit: Days of therapy
Arm/Group | Endoscopic Release | Standard Open Release
Number analyzed (Participants) | 12 | 13
Days of therapy | 3.9 (3.7) | 5.7 (5.7)
Statistical Analysis 1: Comparison: Endoscopic Release vs Standard Open Release; Test type: Other; p = 0.748, Wilcoxon (Mann-Whitney)

5. Secondary Outcome: Pain Medication Use
Description: Number of days opiates used after surgery
Time Frame: End of Study (6 months after treatment)
Population: All available values included in analysis.
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Endoscopic Release | Standard Open Release
Number analyzed (Participants) | 12 | 13
Days | 0 (0) | 0.3 (0.8)
Statistical Analysis 1: Comparison: Endoscopic Release vs Standard Open Release; Test type: Other; p = 0.184, Wilcoxon (Mann-Whitney)

6. Secondary Outcome: Number of Complications
Description: Injury to tendons, nerves, or digital vessels, surgical site dehiscence or surgical site infections requiring antibiotics
Time Frame: Through study completion, an average 1 year
Measure: Number; unit: Complications
Arm/Group | Endoscopic Release | Standard Open Release
Number analyzed (Participants) | 13 | 13
Complications | 0 | 1
Statistical Analysis 1: Comparison: Endoscopic Release vs Standard Open Release; Test type: Other; p = 0.382, Chi-squared

7. Secondary Outcome: Rate of Recurrence
Description: Triggering of treated finger, confirmed on physical exam by treating physician, requiring re-operation
Time Frame: At any time point after treatment; through study completion, an average 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | Endoscopic Release | Standard Open Release
Number analyzed (Participants) | 13 | 13
Participants | 0 | 1
Statistical Analysis 1: Comparison: Endoscopic Release vs Standard Open Release; Test type: Other; p = 0.382, Chi-squared

ADVERSE EVENTS:
Time Frame: Through study completion, an average 1 year
Arm/Group | Endoscopic Release | Standard Open Release
All-Cause Mortality (participants affected / at risk) | 1/13 | 0/13
Serious Adverse Events (participants affected / at risk) | 0/13 | 0/13
Other Adverse Events (participants affected / at risk) | 0/13 | 0/13

LIMITATIONS AND CAVEATS:
Lack of randomization and blinding.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-12-01): https://cdn.clinicaltrials.gov/large-docs/77/NCT03883477/Prot_SAP_000.pdf